CLINICAL TRIAL: NCT02466698
Title: A Feasibility Randomized Trial of Intestinal Lavage for the Treatment of Severe C. Difficile Infections
Brief Title: Intestinal Lavage for the Treatment of Severe C. Difficile Infections
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Tina Mele, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 106184
Record Dates: First submitted 2015-06-04; First posted 2015-06-09 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Clostridium Difficile
Keywords: Colectomy; Surgical Procedures, Operative
MeSH Terms: interventions — polyethylene glycol 3350; Vancomycin; Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intestinal Lavage (Experimental): A nasojejunal tube and fecal management system will be inserted. Intestinal lavage with PEG is initiated and increased to a goal rate of 400cc/hour to a total of 8L of PEG. In the absence of an ileus, lavage should be initiated at 200cc/hr. Tolerance is confirmed if the rectal effluent volume is ≥50% of the lavage volume over the first 6 hours and no emesis has developed. If the consulting surgical service suspects a significant ileus, the lavage is initiated at 100cc/hr. If tolerance is confirmed the lavage rate is increased in a stepwise fashion. Antibiotic regimen will consist of Vancomycin 500mg via nasojejunal every 6 hours and Metronidazole 500 mg IV three times daily for 14 days. PEG will be held for 2 hours after administration of Vancomycin.
  Interventions: Procedure: Intestinal Lavage; Drug: Vancomycin; Drug: PEG; Drug: Metronidazole
- Usual Care (Active Comparator): Patients will receive usual care for severe CDI. This includes an antibiotic regimen of Vancomycin 500mg orally every 6 hours and Metronidazole 500mg IV three times daily for 14 days. The usual care group will receive the same antibiotic doses as the experimental arm of the study. For both arms, indications to escalate treatment to surgical intervention will ultimately be based on the clinical assessment by the surgical service. An absolute indication for surgery is perforation. Other indications such as toxic megacolon, worsening peritonitis or biochemical profile lavage are relative indications that vary according to clinician and individual patient characteristics.
  Interventions: Drug: Vancomycin; Drug: Metronidazole

INTERVENTIONS:
Procedure: Intestinal Lavage — A nasojejunal tube and fecal management system will be inserted. Intestinal lavage with PEG is initiated and increased to a goal rate of 400cc/hour to a total of 8L of PEG. In the absence of an ileus, lavage should be initiated at 200cc/hr. Tolerance is confirmed if the rectal effluent volume is ≥50% of the lavage volume over the first 6 hours and no emesis has developed. If the consulting surgical service suspects a significant ileus, the lavage is initiated at 100cc/hr. If tolerance is confirmed the lavage rate is increased in a stepwise fashion. Antibiotic regimen will consist of Vancomycin 500mg via nasojejunal every 6 hours and Metronidazole 500 mg IV three times daily for 14 days. PEG will be held for 2 hours after administration of Vancomycin.
  Other Names: PEG Lavage
  Arms: Intestinal Lavage
Drug: Vancomycin — Patients will receive standard antibiotic treatment for severe CDI. This includes an antibiotic regimen of Vancomycin 500mg orally every 6 hours and Metronidazole 500mg IV three times daily for 14 days. The standard medical care group (active comparator group) will receive the same antibiotic doses as the experimental arm of the study For both arms, indications to escalate treatment to surgical intervention will ultimately be based on the clinical assessment by the surgical service. An absolute indication for surgery is perforation. Other indications such as toxic megacolon, worsening peritonitis or biochemical profile lavage are relative indications that vary according to clinician and individual patient characteristics.
  Other Names: Antibiotic-V
Drug: PEG — Polyethylene glycol 3350, 8L in 48 hours, via a nasojejunal tube will be used to facilitate intestinal lavage.
  Other Names: Polyethylene glycol 3350
  Arms: Intestinal Lavage
Drug: Metronidazole — Patients will receive standard antibiotic treatment for severe CDI. This includes an antibiotic regimen of Vancomycin 500mg orally every 6 hours and Metronidazole 500mg IV three times daily for 14 days. The standard medical care group (active comparator group) will receive the same antibiotic doses as the experimental arm of the study For both arms, indications to escalate treatment to surgical intervention will ultimately be based on the clinical assessment by the surgical service. An absolute indication for surgery is perforation. Other indications such as toxic megacolon, worsening peritonitis or biochemical profile lavage are relative indications that vary according to clinician and individual patient characteristics.
  Other Names: Antibiotic-M

SUMMARY:
Clostridium Difficile infections (CDIs) are treated initially with antibiotic therapy and supportive care, with surgical intervention reserved for patients with significant systemic toxicity or perforation. Severe CDI may be refractory to medical management and require surgical intervention, carrying a mortality of approximately 40%.

Mortality associated with CDI increases significantly as the severity of the infection increases. In patients failing medical management, earlier operation is associated with decreased mortality. However, the lack of validated tools to predict the necessity for surgical intervention, combined with the significant morbidity associated with total colectomy significantly reduces the likelihood of patients receiving early surgical intervention. The purpose of the proposed study is to assess the addition of intestinal PEG lavage via nasojejunal tube to usual care in the treatment of adult patients with severe CDI who have no immediate indication for surgical intervention.

DETAILED DESCRIPTION:
Despite a lack of definitive evidence, total abdominal colectomy (TAC) is currently recommended as the surgical intervention of choice in the setting of severe-complicated CDI. This recommendation was based on meta-analysis of studies comparing TAC to partial colectomy or other surgery (such as exploratory laparotomy without colectomy, or ostomy formation) or no surgery, which did not find any statistical mortality difference. This recommendation is based on the results of sensitivity analysis and an expert panel consensus that considered the potential for confounding factors such as TAC occurring later in the course of the disease and on sicker patients, and on anticipated patient values that would pace value on a definitive procedure being the initial surgical intervention.

Given the high mortality of fulminant CDI, early surgical intervention is recommended. However, data regarding the optimal timing for surgical intervention is lacking. Meta-analyses and guidelines strongly recommend early surgical management, defined as being before the development of shock or the requirement for vasopressors, based on very low quality evidence, but with the potential for significant mortality reduction.

On the basis of CDI being a toxin mediated inflammatory process of the colonic mucosa, Neal et al hypothesized that surgical diversion of the fecal stream with a loop ileostomy and intraoperative antegrade colonic lavage may effectively treat severe CDI. Widely referred to as the 'Pittsburgh Protocol,' the regimen included colonic lavage with 8 litres of polyethylene glycol (PEG 3350) intra-operatively after formation of a loop ileostomy, followed by antegrade Vancomycin flushes (500mg in 500cc Ringer's Lactate TID) and IV Metronidazole (500mg TID) for 10 days. The study utilized a before-and-after methodology comparing the experimental protocol to historical controls. Forty-two patients were submitted to the regimen over 18 months. Three patients required reoperation for TAC. 30-day mortality was 19% in the intervention cohort, compared to 50% in the control. 79% of survivors went on to ileostomy reversal within 6 months of surgery. One of the potential benefits of this regimen is that given the reduced morbidity compared to TAC, practitioners may have been offering surgical intervention earlier in the management of CDI and not exclusively as a therapy of last resort. Despite the limited sample size and methodological shortcoming of this study, this treatment regime has been adopted in some centres for select cases. A randomized controlled trial to compare this less invasive surgical approach with total abdominal colectomy was closed prematurely given lack of meaningful patient enrolment (clinicaltrials.gov identifier NCT01441271).

Given the positive results of fecal diversion and antegrade lavage and vancomycin flushed proposed by Neal et al, combined with the limited data regarding the benefit of intracolonic vancomycin, a novel treatment was instituted at London Health Sciences Centre (LHSC) to accomplish lavage of the colon and vancomycin flushes in an antegrade fashion using a nasojejunal feeding tube to facilitate delivery in select patients. The protocol allows for lavage and intracolonic antibiotic delivery similar to that provided by the 'Pittsburgh protocol' without surgical fecal diversion.

A small preliminary cohort of patients completing this protocol at LHSC is being assessed retrospectively, comparing outcomes to a group undergoing the Pittsburgh protocol and initial total colectomy. The study was approved by the Western University Research Ethics Board (REB File # 104944). Interim analysis of the past 24 months includes 13 patients undergoing the study protocol, 9 undergoing the Pittsburgh protocol and 17 undergoing initial colectomy. Despite significant limitations of the study methodology, the results are encouraging and further study is warranted, especially given the significant mortality associated with fulminant CDI.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>= 18 years) inpatients at LHSC with symptomatic CDI (diarrhea or colonic ileus)
* CDI confirmed by standard hospital microbiology lab testing
* Patients must meet criteria for severe CDI, defined as either: white blood cell > 15,000 or Serum Creatinine > 1.5 times the pre-morbid level
* Patients must have at least one additional risk factor for severity:

  i. Fever >38.5 (if no other source of fever suspected) ii. Vasopressor requirement iii. Mechanical ventilation requirement iv. Serum lactate >5 mmol/L v. Colonic distension (>6cm transverse colon diameter on abdominal Xray or CT) vi. Colonic wall thickening, on abdominal Xray or CT, as reported by radiology. vii. Calculated ATLAS score ≥ 4

Exclusion Criteria:

* The patient is deemed to have an immediate indication for surgery related to the diagnosis of CDI by the on call General Surgery service.
* Pre-existing bowel discontinuity (e.g. ileostomy).
* General Surgery service or most responsible care team deem the patient to have a contraindication to nasojejunal tube or fecal management system
* Patients anticipated to be intolerant of the study regimen (e.g. severe ileus, unable to tolerate oral intake, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Number of eligible participants recruited into the study | 12 months
  Recruited participants

SECONDARY OUTCOMES:
Number of participants meeting study inclusion criteria | 12 months
  Included participants
Number of participants who complete the assigned study protocol | 12 months
  Completed study participants
Number of participants who complete the treatment protocol without an adverse event | 12 months
  Participants with no adverse events
Number of participants with a complication or adverse event | 12 months
  Participants with adverse events
Number of participants who require initiation of mechanical ventilation following protocol initiation | 12 months
  Participants requiring mechanical ventilation
Number of participants who require operative intervention for CDI treatment | 12 months
  Participants requiring operative intervention
Surgeons' indication for operative intervention | 12 months
  Surgeons will indicate the indication for operative intervention for any patient that is taken to the operating theatre for CDI treatment
30-day all-cause mortality | 12 months
  Mortality within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Tina E Mele, MD PhD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-dentified data available upon reasonable request after publication of study results
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing after publishing the study.
Access Criteria: A direct request from PI.

REFERENCES:
- [Derived] McCreery G, Jones PM, Kidane B, DeMelo V, Mele T; ERASE C. difficile (Early Rescue from Acute SEvere Clostridium difficile) Trials Group. Polyethylene glycol intestinal lavage in addition to usual antibiotic treatment for severe Clostridium difficile colitis: a randomised controlled pilot study. BMJ Open. 2017 Jul 31;7(7):e016803. doi: 10.1136/bmjopen-2017-016803. PMID 28760801